CLINICAL TRIAL: NCT00004862
Title: A Phase I Study of G3139 (NSC 683428) in Combination With Salvage Chemotherapy for Treatment of Refractory and Relapsed Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (ALL)
Brief Title: Augmerosen Plus Fludarabine and Cytarabine in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01399; OSU-99H0257; OSU-9977; NCI-T99-0057; CDR0000067515 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-03-07; First posted 2004-01-29 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2002-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; oblimersen; Cytarabine; fludarabine phosphate

ARMS (1):
- Arm I (Experimental): Patients receive augmerosen IV continuously on days 1-10 and filgrastim (G-CSF) subcutaneously beginning on day 5 and continuing until blood counts recover. Patients receive fludarabine IV over 30 minutes followed 3.5 hours later by cytarabine IV over 4 hours on days 6-10. Patients who achieve complete response (CR) receive a second course beginning 4 weeks after completion of the first course. Patients who achieve CR and have a matched sibling or unrelated bone marrow donor may undergo allogeneic bone marrow transplantation. Cohorts of 3-6 patients receive escalating doses of fludarabine and cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Biological: filgrastim; Biological: oblimersen sodium; Drug: cytarabine; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: filgrastim
Biological: oblimersen sodium
Drug: cytarabine
Drug: fludarabine phosphate

SUMMARY:
Phase I trial to study the effectiveness of augmerosen plus fludarabine and cytarabine in treating patients who have refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Gene therapy such as augmerosen may make cancer cells more sensitive to chemotherapy drugs. Combining more than one drug with augmerosen may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of fludarabine and cytarabine when combined with augmerosen (G3139) in patients with refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia and recommend a starting dose for phase II studies.

II. Determine the qualitative and quantitative toxic effects of this regimen in these patients with regard to organ specificity, time course, predictability, and reversibility.

III. Document the therapeutic response in patients treated with this regimen. IV. Measure bcl-2 and related antiapoptotic and proapoptotic proteins in circulating and/or marrow leukemia cells before, during, and after treatment with G3139.

V. Measure WT1 expression in leukemic blasts as a surrogate marker for minimal residual disease and correlate it with bcl-2 and related antiapoptotic and proapoptotic gene expression.

VI. Determine the time required for bcl-2 levels to recover after treatment with this regimen.

VII. Determine if TP53 mutations are present in leukemic blasts and how these mutations may affect expression of BAX, level of treatment induced apoptosis, and clinical endpoints.

VIII. Assess apoptosis in leukemic cells before, during, and after treatment with this regimen.

IX. Determine the pharmacokinetics of fludarabine and cytarabine in patients treated with this regimen.

X. Perform pharmacodynamic studies of fludarabine and cytarabine on the leukemic cells of patients prior to treatment.

OUTLINE: This is a dose-escalation study of fludarabine and cytarabine.

Patients receive augmerosen IV continuously on days 1-10 and filgrastim (G-CSF) subcutaneously beginning on day 5 and continuing until blood counts recover. Patients receive fludarabine IV over 30 minutes followed 3.5 hours later by cytarabine IV over 4 hours on days 6-10. Patients who achieve complete response (CR) receive a second course beginning 4 weeks after completion of the first course. Patients who achieve CR and have a matched sibling or unrelated bone marrow donor may undergo allogeneic bone marrow transplantation. Cohorts of 3-6 patients receive escalating doses of fludarabine and cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia
* Marrow cellularity must be at least 20%
* Must have diagnostic lumbar puncture and treatment with prophylactic intrathecal methotrexate within 1 week prior to entering study
* No active CNS involvement
* CNS involvement allowed if no residual leukemic cells are detected in CSF following intrathecal chemotherapy

PATIENT CHARACTERISTICS:

* Age: 16 and over
* Performance status: ECOG 0-2
* Life expectancy: At least 4 weeks
* Bilirubin no greater than 2 times upper limit of normal(ULN)

  * ALT and AST no greater than 2 times ULN
  * Alkaline phosphatase no greater than 2 times ULN*
  * Unless attributable to malignancy
* Creatinine no greater than 1.5 mg/dL unless attributable to malignancy
* No symptomatic congestive heart failure
* No unstable angina pectoris No or cardiac arrhythmia
* Resting cardiac ejection fraction no less than 45% unless attributable to malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before and during study
* No history of allergy to study medications
* No uncontrolled concurrent illness
* No active infection
* No serious medical or psychiatric illness that would preclude informed consent or limit survival to less than 4 weeks

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior chemotherapy except hydroxyurea
* No concurrent corticosteroids except for grade 4 toxicity unresponsive to all other agents
* At least 4 weeks since prior radiotherapy
* No other concurrent investigational or standard agents or therapies for leukemia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1999-10; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States